CLINICAL TRIAL: NCT01564641
Title: A Prospective, Multicenter Study of the ConforMIS iDuo(R) G2 Bicompartmental Knee Repair System
Brief Title: Study of the ConforMIS iDuo(R) G2
Status: Terminated | Type: Observational
Why Stopped: Decision of investigational team
Sponsor: Restor3D (Industry)
Responsible Party: Sponsor
Other Study IDs: 11-001
Record Dates: First submitted 2012-03-12; First posted 2012-03-28 (Estimated); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Bicompartmental Osteoarthritis
Keywords: knee; osteoarthritis; bicompartmental; arthroplasty; joint diseases
MeSH Terms: conditions — Osteoarthritis; Joint Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- iDuo G2: iDuo G2 to be implanted in the patient.
  Interventions: Device: iDuo G2

INTERVENTIONS:
Device: iDuo G2 — single comparator

SUMMARY:
To evaluate the ConforMIS iDuo G2 implant

DETAILED DESCRIPTION:
This is a prospective, multicenter study. The investigators will be evaluating the ConforMIS iDuo G2 implant.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical condition included in the approved Indications For Use for the iDuo® G2
2. Bicompartmental osteoarthritis defined as Medial and patellofemoral osteoarthritis, or Lateral and patellofemoral arthritis as confirmed by the investigator's assessment of disease status at screening visit. Disease status is assessed by Clinical and Radiographic assessment. In addition, CT arthrogram assessment may be utilized for diagnosis.
3. Willingness to participate in the clinical study, to give informed consent and to attend all follow-up visits
4. > 18 years of age

Exclusion Criteria:

1. BMI > 40
2. Active malignancy (defined as a history of any invasive malignancy - except non-melanoma skin cancer), unless patient has been treated with curative intent and there have been no clinical signs or symptoms of the malignancy for at least 5 years
3. Poorly controlled diabetes
4. Neuromuscular conditions which prevent patient from participating in study activities
5. Active local or systemic infection
6. Immunocompromised
7. Fibromyalgia or other general body pain related condition
8. Rheumatoid arthritis or other forms of inflammatory joint disease
9. Loss of bone or musculature, osteonecrosis, neuromuscular or vascular compromise in the area of the joint to be operated to an extent that the procedure is unjustified
10. Diagnosed or receiving treatment for Osteoporosis
11. Other physical disability affecting the hips, spine, or contralateral knee
12. Severe instability due to advanced loss of osteochondral structure
13. Prior arthroplasty of the affected knee
14. Compromised ACL, PCL or collateral ligament
15. Severe fixed valgus or varus deformity of >15º
16. Extensor lag > 15 º
17. Fixed flexion contracture ≥ 10 º
18. Prior history of failed implant surgery of the joint to be treated, including high tibial osteotomy (HTO)
19. Unwilling or unable to comply with study requirements
20. Participation in another clinical study which would confound results
21. If during intra-op, it is noted that the patient has tri-compartmental disease, then the patient is considered a screen fail

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting this specific form of osteoarthritis at participating sites with IRB approval.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2012-05 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2022-11-18 (Actual)

PRIMARY OUTCOMES:
Pain and function | 3 months
  By using questionnaires, we will look at pain and function scores at this time point

SECONDARY OUTCOMES:
Pain and function at follow up time points | 1, 2, 5 and 10 years post implant
  By using questionnaires, we will look at pain and function scores at these time points
Revision rates | Patient will be observed for 10 years post implant
  Capture revision rates
Incidence of major procedure related and device related complications | Patient will be observed for 10 years post implant
  To capture any procedure or device related complications
Post operative limb alignment | X rays will be taken at 1 year, 2 year, 5 year and 10 year follow ups
Radiographic implant position | X rays will be taken at 1 year, 2 year, 5 year and 10 year follow ups
Radiographic loosening, radiolucencies | X rays will be taken at 1 year, 2 year, 5 year and 10 year follow ups
Length of procedure | Day of surgery
  Timing from skin to cement
Length of hospital stay | Patient will be followed from admission to discharge with an average of about 5 days
  measure length of stay from admission to discharge
Blood loss during surgery | Day of surgery
Intraoperative blood replacement volume | Day of surgery

CONTACTS AND LOCATIONS:
Overall Officials: L Rolston, MD, Principal Investigator — Forest Ridge
Locations (3):
- United States (3):
  - Forest Ridge Medical Pavilion, New Castle, Indiana
  - Ochsner Sports Medicine Institute, New Orleans, Louisiana
  - Mansfield Orthopaedics, Morrisville, Vermont

IPD SHARING:
Plan to Share IPD: No